CLINICAL TRIAL: NCT02501200
Title: Clinical Trial to Assess the Pharmacokinetic Characteristics and Safety/Tolerability of CKD-391 in Healthy Male Subjects
Brief Title: CKD-391 Pharmacokinetic Study Phase I
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 152BE15026
Record Dates: First submitted 2015-07-16; First posted 2015-07-17 (Estimated); Last update posted 2016-12-26 (Estimated); Status verified 2015-10

CONDITIONS: Healthy
Keywords: Dyslipidemia; CKD-391; Atorvastatin; Ezetimibe
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TR group (Experimental): CKD-391 and combination dose of Atrovastatin and Ezetimibe in order
  Interventions: Drug: CKD-391; Drug: Atrovastatin and Ezetimibe combination therapy
- RT group (Experimental): combination dose of Atrovastatin and Ezetimibe and CKD-391 in order
  Interventions: Drug: CKD-391; Drug: Atrovastatin and Ezetimibe combination therapy

INTERVENTIONS:
Drug: CKD-391 — Investigational product is prescribed to all of randomized subjects for two times.
Drug: Atrovastatin and Ezetimibe combination therapy — Investigational products are prescribed to all of radomized subjects for two times.

SUMMARY:
A randomized, open-label, 2-way crossover study to compare the pharmacokinetics and safety CKD-391 to coadministration Atorvastatin and Ezetimibe in health volunteers.

DETAILED DESCRIPTION:
To compare the CKD-391 (Experimental product) to the dose Atorvastatin calcium and Ezetimibe combination in health male subjects is the purpose of this trial.

Following are evaluated in this trial; Characteristics and safety/Tolerability Of CKD-391.

ELIGIBILITY:
Inclusion Criteria:

* Bwt >=50kg, BMI 18.5~25
* signed the informed consent form prior to the study participation

Exclusion Criteria:

* - Clinically significant disease
* Subject has signs of symptoms of acute disease within 28 days of starting administration of investigational drug
* Clinically significant allergic disease
* Impossible to taking the institutional standard meal
* Previously donate whole blood within 60 days or component blood within 20 days
* Previously participated in other trial within 90 days
* Continued to be taking caffeine (caffeine > 5 cup/day), drinking(alcohol > 30 g/day) or cannot stop drinking or severe heavy smoker(cigarette > 10 cigarettes per day)during clinical trials
* An impossible one who participates in clinical trial by investigator's decision including laboratory test result

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2015-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
AUClast | up to 96 hours post dose
Cmax | up to 96 hours post dose

SECONDARY OUTCOMES:
Tmax | up to 96 hours post dose
T1/2 | up to 96 hours post dose
AUCinf | up to 96 hours post dose
Adverse events | up to 24days post dose

CONTACTS AND LOCATIONS:
Overall Officials: Choon Ok Kim, Ph.D, Principal Investigator — Severance Hospital

IPD SHARING:
Plan to Share IPD: No